CLINICAL TRIAL: NCT03305510
Title: Prospective Cohort Study About Vitamin D Deficiency of Couples and Infertility
Brief Title: Vitamin D Deficiency of Couples and Infertility
Status: Completed | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Liu Jiang, MD, Tongji Hospital
Other Study IDs: Reproductive center of Tongji
Record Dates: First submitted 2017-10-08; First posted 2017-10-10 (Actual); Last update posted 2017-10-10 (Actual); Status verified 2017-10

CONDITIONS: Vitamin D Deficiency; Infertility; Couples; In-vitro Fertilization
MeSH Terms: conditions — Vitamin D Deficiency; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Vitamin D deficiency: The level of vitamin D is below 20ng/ml.
  Interventions: Diagnostic Test: vitamin D is below 20ng/ml
- Vitamin D insufficient: The level of vitamin D is between 20ng/ml and 30ng/ml.
- Vitamin D sufficient: The level of vitamin D is above 30ng/ml.

INTERVENTIONS:
Diagnostic Test: vitamin D is below 20ng/ml
  Groups: Vitamin D deficiency

SUMMARY:
Between March 2016 and March 2017, we performed a large retrospective, non-interventional, single-center cohort study and measured 25(OH)D3 plasma levels prior to ovarian stimulation in couples who underwent IVF/ICSI.And we analysed the correlation of vitamin D status and reproductive capacity .

DETAILED DESCRIPTION:
Before conducting ovarian stimulation, all couples must conduct preoperative routine examination such as routine blood test, blood group examination and infectious disease examination. We collected 2ml remaining blood from the examination by use of sodium heparin, which then conducted 1,25(OH)2D3 assay by liquid chromatography-tandem mass spectrometry.

All patients underwent a standardized ovarian stimulation regimen, oocyte retrieval, and fertilization, followed by a planned fresh or frozen embryo transfer.Normal fertilization rate was defined as the presence of two pronuclei (2PN) at the time of fertilization assessment, 16-19 h after ICSI or conventional insemination. The percentage of top quality embryos was defined as the percentage of top quality embryos among the total number of 2PN embryos. Blastocyst forming rate was calculated as number of formed blastocysts devided by number of cultured blastocysts.

ELIGIBILITY:
Inclusion Criteria:

* couples who underwent IVF/ICSI.

Exclusion Criteria:

* sperm or egg donation, PGD or PGS,TESA or PESA, ovum frozen ,no oocyte for fertilization.

Ages: 20 Years to 42 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: non-interventional, single-center cohort study and measured 25(OH) D plasma levels prior to ovarian stimulation in couples who underwent IVF/ICSI.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
fertilization rate | the time of fertilization assessment, 16-19 hours after ICSI or conventional insemination
  Normal fertilization rate was defined as the presence of two pronuclei (2PN) at the time of fertilization assessment, 16-19 h after ICSI or conventional insemination. The percentage of top quality embryos was defined as the percentage of top quality embryos among the total number of 2PN embryos. Blastocyst forming rate was calculated as number of formed blastocysts devided by number of cultured blastocysts.

CONTACTS AND LOCATIONS:
Overall Officials: Kun Qian, Doctor, Study Chair — Tongji Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jiang L, Yang J, Song J, Hu Y, Qian K. Normal fertilisation rates and serum 25-OHD levels among couples undergoing in-vitro fertilisation: a prospective cohort study. BMC Pregnancy Childbirth. 2020 Jun 5;20(1):346. doi: 10.1186/s12884-020-02959-z. PMID 32503520